CLINICAL TRIAL: NCT02767674
Title: Phase III,Randomized Controlled Trial of R-GemOx Versus R-miniCHOP Regimen in First-line Treatment of Elderly Diffuse Large B Cell Lymphoma
Brief Title: Trial of R-GemOx Versus R-miniCHOP Regimen in First-line Treatment of Elderly Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JSPH-002
Record Dates: First submitted 2016-05-07; First posted 2016-05-10 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: R-Gemox; R-miniCHOP; elderly patients with diffuse large B cell lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Gemcitabine; Oxaliplatin; Cyclophosphamide; Vindesine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-GemOx (Experimental): Rituximab: 375 mg/m2 IV day0, Gemcitabine 1g/m2 IV day 1, oxaliplatin 100mg/m2 IV day1(every 14 days)
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin
- R-miniCHOP (Active Comparator): Rituximab, 375 mg/m2 IV d0 Cyclophosphamide 400 mg/m2 IV d1 Epirubicin 35 mg/m2 IV d1 vindesine 2 mg IVP d1 Prednisone 40mg/m2 PO d1-5(every 21 days a cycle)
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Epirubicin Injectable Product; Drug: Vindesine; Drug: Prednisone

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 IVD day0
Drug: Gemcitabine — Gemcitabine 1 g/m2 IVD day 1
  Arms: R-GemOx
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 IVD day1
  Arms: R-GemOx
Drug: Cyclophosphamide — Cyclophosphamide 400 mg/m2 IVD d1
  Arms: R-miniCHOP
Drug: Epirubicin Injectable Product — Epirubicin 35 mg/m2 IVD d1
  Arms: R-miniCHOP
Drug: Vindesine — Vindesine 2 mg IVP d1
  Arms: R-miniCHOP
Drug: Prednisone — Prednisone 40mg/m2 PO d1-5
  Arms: R-miniCHOP

SUMMARY:
The purpose of this study is to investigate efficacy and safety of R-GemOx Versus R-miniCHOP as first-line treatment of elderly patients with Diffuse large B cell lymphoma

DETAILED DESCRIPTION:
Gemcitabine and Oxaliplatin(GemOx) shows effective activity in patients with relapsed diffuse large-cell lymphoma and other solid tumors. Our Previous study showed that two-weekly regimen of rituximab combined with GemOx regimen acheived comparable response rate to R-miniCHOP.The investigators therefore design this open-label,phase III and random trial to compared the safety and efficacy of R-Gemox versus R-miniCHOP as first-line treatment of elderly patients with diffuse large B cell lymphoma.

Primary Outcome Measures:

• 2-year overall survival rate

Secondary Outcome Measures:

* 2-year progression free survival rate
* overall response rate
* safety and toxicity Enrollment:258 Study Start Date: June 2016 Primary Completion Date: June 2019

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diffuse large B cell lymphoma（With exception of Primary mediastinal large B cell lymphoma、Primary central nervous system lymphoma、HIV-related lymphoma);
2. New-diagnosed and untreated;
3. Age older than 80 years or older than 70 years with ECOG PS ≥ 2;
4. Ann Arbor stage I to stage IV disease;
5. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Poor hepatic and/or renal function, defined as total bilirubin, ALT, AST, Cr more than two fold of upper normal level, unless these abnormalities were related to the lymphoma;
2. Poor bone-marrow reserve, defined as neutrophil count less than 1.5×10⁹/L or platelet count less than 75×10⁹/L, unless caused by bone marrow infiltration;
3. Presence of Grade III nervous toxicity with two weeks;
4. New York Heart Association class III or IV cardiac failure; or Ejection fraction less than 50%;or history of following disease in past 6 months: acute coronary syndrome、acute heart failure、severe ventricular arrhythmia
5. Positive HIV, syphilis,HCV, or HBV virus load(HBV DNA)> 1×10'4copies/ml;
6. CNS or meningeal involvement;
7. Concomitant malignancy other than aggressive B cell lymphoma and need to Treat, with the exception of non-melanoma skin tumours or stage 0 (in situ) cervical carcinoma,or history of cancer more than 5 years;
8. Concomitant with other hematologic diseases(such as leukemia, hemophilia primary myelofibrosis) which investigator it unsuitable to be enrolled into this clinical trial;
9. Active and severe infectious diseases;
10. Major surgery within three weeks;
11. Any potential drug abuse, medical, psychological or social conditions which may disturb this investigation and assessment.
12. In any conditions which investigator considered ineligible for this study.
13. Known sensitivity or allergy to investigational Product.

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2016-05; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival rate | One year
  from the date of inclusion to date of death, irrespective of cause

SECONDARY OUTCOMES:
2-year progression free survival rate | One year
  from date of inclusion to date of progression, relapse, or death from any causePFS：from date of inclusion to date of progression, relapse, or death from any cause
overall response rate | One year
  overall response rate after treated by R-GemOx or R-miniCHOP overall response rate after treated by R-GemOx or R-miniCHOP regimen

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D., Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (6):
- China (6):
  - Tongji Medical College of HUST, Wuhan, Hubei
  - The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital), Nanjing, Jiangsu
  - QiLu Hospital of Shandong University, Jinan, Shandong
  - Shandong Province Hospital, Jinan, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Sudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Result] Oyama T, Yamamoto K, Asano N, Oshiro A, Suzuki R, Kagami Y, Morishima Y, Takeuchi K, Izumo T, Mori S, Ohshima K, Suzumiya J, Nakamura N, Abe M, Ichimura K, Sato Y, Yoshino T, Naoe T, Shimoyama Y, Kamiya Y, Kinoshita T, Nakamura S. Age-related EBV-associated B-cell lymphoproliferative disorders constitute a distinct clinicopathologic group: a study of 96 patients. Clin Cancer Res. 2007 Sep 1;13(17):5124-32. doi: 10.1158/1078-0432.CCR-06-2823. PMID 17785567
- [Result] Peyrade F, Jardin F, Thieblemont C, Thyss A, Emile JF, Castaigne S, Coiffier B, Haioun C, Bologna S, Fitoussi O, Lepeu G, Fruchart C, Bordessoule D, Blanc M, Delarue R, Janvier M, Salles B, Andre M, Fournier M, Gaulard P, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte (GELA) investigators. Attenuated immunochemotherapy regimen (R-miniCHOP) in elderly patients older than 80 years with diffuse large B-cell lymphoma: a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2011 May;12(5):460-8. doi: 10.1016/S1470-2045(11)70069-9. Epub 2011 Apr 7. PMID 21482186
- [Result] Lopez A, Gutierrez A, Palacios A, Blancas I, Navarrete M, Morey M, Perello A, Alarcon J, Martinez J, Rodriguez J. GEMOX-R regimen is a highly effective salvage regimen in patients with refractory/relapsing diffuse large-cell lymphoma: a phase II study. Eur J Haematol. 2008 Feb;80(2):127-32. doi: 10.1111/j.1600-0609.2007.00996.x. Epub 2007 Nov 20. PMID 18005385
- [Result] Cabanillas F. Rituximab in DLBCL: 6 years on. Lancet Oncol. 2011 Oct;12(11):984-5. doi: 10.1016/S1470-2045(11)70251-0. Epub 2011 Sep 21. No abstract available. PMID 21940215
- [Result] Park S, Lee J, Ko YH, Han A, Jun HJ, Lee SC, Hwang IG, Park YH, Ahn JS, Jung CW, Kim K, Ahn YC, Kang WK, Park K, Kim WS. The impact of Epstein-Barr virus status on clinical outcome in diffuse large B-cell lymphoma. Blood. 2007 Aug 1;110(3):972-8. doi: 10.1182/blood-2007-01-067769. Epub 2007 Mar 30. PMID 17400912